CLINICAL TRIAL: NCT03844646
Title: Real-Time Continuous Glucose Monitoring to Aid Weight Loss in Prediabetes
Brief Title: Continuous Glucose Monitoring to Aid Weight Loss in Prediabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sun H Kim, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49402; P30DK116074 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Weight Loss; PreDiabetes
MeSH Terms: conditions — Weight Loss; Prediabetic State | interventions — Nutritionists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CGM plus dietitian (Experimental): Intermittent use of a continuous glucose monitor (CGM) plus dietitian support
  Interventions: Device: CGM; Other: Dietitian
- Dietitian only (Other): Dietitian support only
  Interventions: Other: Dietitian

INTERVENTIONS:
Device: CGM — Intermittent use of a continuous glucose monitor (CGM)
  Arms: CGM plus dietitian
Other: Dietitian — Monthly meetings with a dietitian

SUMMARY:
The primary objective of this study is to determine whether intermittent use of continuous glucose monitor will facilitate weight loss in individuals who are overweight/obese with prediabetes.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) has revolutionized the treatment of patients on intensive insulin therapy and its utility can also be harnessed to help individuals with prediabetes make healthful lifestyle changes. Successful weight loss requires adherence to lower calories, regular exercise, and self-monitoring. This proposal will test the hypothesis that intermittent CGM will facilitate all of these components for successful weight loss by functioning as a continuous self-monitor and guiding healthful food choices and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese (BMI 25-40 kg/m2)
* Prediabetes (fasting glucose 100-125 mg/dL and/or HbA1c 5.7-6.4%)

Exclusion Criteria:

* On glucose-lowering medications (e.g., metformin)
* On weight-loss medications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Kim, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CGM Plus Dietitian: Intermittent use of a continuous glucose monitor (CGM) plus monthly support meetings with a dietitian.
- Dietitian Only: Monthly support meetings with a dietitian.
Period: Overall Study
Arm/Group | CGM Plus Dietitian | Dietitian Only
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGM Plus Dietitian | Dietitian Only | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 2 | 5
  Hispanic | 2 | 0 | 2
  NonHispanic White | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Amount of Weight Lost (kg)
Description: Weight lost during the study
Time Frame: Baseline to end of study (3 months)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | CGM Plus Dietitian | Dietitian Only
Number analyzed (Participants) | 8 | 4
kg
  Baseline | 77.4 (8.4) | 74.9 (7.5)
  Change at month 3 | -2.9 (4.0) | -3.1 (0.6)

2. Secondary Outcome: Number of Participants Reporting at Least 5 Days of Moderate Physical Activity of 30 Minutes or More
Time Frame: Baseline to end of study (3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Plus Dietitian | Dietitian Only
Number analyzed (Participants) | 8 | 4
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | CGM Plus Dietitian | Dietitian Only
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4

LIMITATIONS AND CAVEATS:
This study did not achieve its planned sample size and is underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03844646/Prot_SAP_001.pdf